CLINICAL TRIAL: NCT04812860
Title: A Multicenter,Randomized, Double-blind, Dose Ranging , Active- and Placebo-controlled, Parallel Groups, Phase II Clinical Trial to Evaluate the Efficacy and Safety of HR18042 Tablets for the Treatment of Postoperative Pain of Impacted Tooth.
Brief Title: A Study to Evaluate the Efficacy and Safety of HR18042 Tablets in the Treatment of Postoperative Pain of Impacted Tooth.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR18042-201
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Moderate to Severe Acute Pain

STUDY DESIGN:
Intervention Model Description: A Multicenter,randomized, double-blind, Dose Ranging , controlled with active treatment and placebo, parallel groups, Phase II clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HR18042 100mg (Experimental)
  Interventions: Drug: HR18042
- HR18042 125mg (Experimental)
  Interventions: Drug: HR18042
- HR18042 200mg (Experimental)
  Interventions: Drug: HR18042
- Tramadol hydrochloride ER 100mg (Active Comparator)
  Interventions: Drug: Tramadol hydrochloride ER
- Placebo to match HR18042 and Tramadol hydrochloride ER (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HR18042 — Tablet, Dosing frequency: once daily, Route of administration: oral
  Arms: HR18042 100mg
Drug: HR18042 — Tablet,Dosing frequency: once daily, Route of administration: oral
  Arms: HR18042 125mg
Drug: HR18042 — Tablet,Dosing frequency: once daily, Route of administration: oral
  Arms: HR18042 200mg
Drug: Tramadol hydrochloride ER — Tablet,Dosing frequency: once daily, Route of administration: oral
  Arms: Tramadol hydrochloride ER 100mg
Drug: Placebo — Tablet,Dosing frequency: once daily, Route of administration: oral
  Arms: Placebo to match HR18042 and Tramadol hydrochloride ER

SUMMARY:
The purpose of this study was to evaluate the Efficacy and safety of HR18042 tablets for the Treatment of Post-surgical Pain After extraction of impacted tooth, find the optimal dose.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old.
2. Subjects must have a plan of extraction of impacted tooth.
3. Subjects with moderate to severe pain (VAS score ≥ 50mm).This must be measured within a maximum of 4 hours after the end of extraction of impacted tooth.
4. weight at least 45kg,and no more than 100kg.
5. If a female is of child-bearing potential, she must be using highly effective methods of contraception throughout the study.
6. Willingness to comply with the study procedures and requirements.
7. willing and able to provide written informed consent for this study.

Exclusion Criteria:

1. any analgesic medication other than preoperative or intraoperative anaesthetic agents within 12h before taking trial medication medication
2. a longacting NSAID within 4 days,or a shortacting NSAID within 1 days prior to dosing.
3. any anti-depressive medication, selective serotonin reuptake inhibitors (SSRIs), diet pills et.al. with 30 days of study entry.
4. Oral surgical site combined with infection.
5. Severe cardiovascular and cerebrovascular diseases.
6. Severe gastrointestinal disease.
7. had a history of seizures or drug or alcohol abuse.
8. uncontrolled hypertension.
9. significant abnormal electrocardiogram
10. significant abnormal laboratory value.
11. Allergic to the study drug and ingredients.
12. Pregnancy, lactation or recent Pregnant plan;
13. Subjects who participated in a clinical research study involving an experimental drug before 30 days of study entry.
14. other conditions unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
the Sum of Pain Intensity Differences（SPID） | 0-8hours
  SPID is derived as the weighted Sum of Pain Intensity Differences (baseline pain - current pain), measured at different time points via the PI-VAS. Time between two consecutive measurements will be used for weighting. Larger values indicate larger pain relief.

SECONDARY OUTCOMES:
the Sum of Pain Intensity Differences（SPID） | 0-4hours
the Sum of Pain Intensity Differences（SPID） | 0-12hours
Pain Intensity Differences（PID） | 0-12hours
  Include pain intensity differences(PIDs) from baseline at each time point. measured at different time points via the PI-VAS.
Pain relief（PAR） | 0-12hours
  pain relief (PAR) on a 5-point Likert scale (0, none, 1, a little, 2, some,3, a lot, 4, complete).
the Sum of Pain relief Differences（SPAR） | 0-4hours
  SPAR is derived as the weighted Sum of Pain relief, measured at different time points via the 5-point Likert scale. Time between two consecutive measurements will be used for weighting. Larger values indicate larger pain relief.
the Sum of Pain relief Differences（SPAR） | 0-8hours
the Sum of Pain relief Differences（SPAR）. | 0-12hours
Subject who reaches a 30% reduction in pain intensity from baseline | 4hours、8hours、12hours
Subject who reaches a 50% reduction in pain intensity from baseline | 4hours、8hours、12hours
time to perceptible pain relief | 0-12hours
time to meaningful pain relief | 0-12hours
  Patients used one stopwatch to record the time to 'perceptible' PAR and another stopwatch for the time to'meaningful' PAR.Patients started timing upon intake of study medication and stopped one stopwatch at the onset of perceptible PAR and another upon achieving meaningful PAR.
Time to first use of rescue medication | 0-12hours
Proportion of subjects who take of at least 1 dose of rescue medication | 0-12hours
Subject's overall assessment of study medication | 12hours
  Patients made an overall assessment of the study medication using a verbal rating scale (excellent, verygood, good, fair, poor).

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Stomatology Sichuan University, Chengdu, Sichuan, China